CLINICAL TRIAL: NCT01570101
Title: Post Market Study - "European Observational Study of the Sapheon™ Closure System for the Definitive Treatment of Incompetent Great Saphenous Veins: A Prospective Single Arm Multicenter Clinical Observational Study"
Brief Title: European Sapheon™ Closure System Observational ProspectivE (eSCOPE) Study
Acronym: eSCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-10763-01
Record Dates: First submitted 2012-03-26; First posted 2012-04-04 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Venous Insufficiency of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CE Marked Sapheon Closure System in GSV (Experimental): CE Marked Sapheon Closure System in closure of incompetent great saphenous veins "GSV" in a routine clinical setting.
  Interventions: Device: CE Marked Sapheon Closure System

INTERVENTIONS:
Device: CE Marked Sapheon Closure System — CE Marked Sapheon Closure System in closure of incompetent great saphenous veins "GSV" in a routine clinical setting.

SUMMARY:
The primary objective for this clinical study is to assess the role of the CE Marked Sapheon Closure System in closure of incompetent great saphenous veins "GSV" in a routine clinical setting.

DETAILED DESCRIPTION:
This is a post market, observational study of closure of the great saphenous vein "GSV". Efficacy and safety (adverse events) will be compared to appropriate literature reports to determine if the results of the treatment of reflux disease with the Sapheon Closure System are consistent with or better than the expectations of the medical community for alternative treatments, specifically Laser Thermal Ablation and Radiofrequency Ablation. Additional comparison points may include measurements of pain and/or length of time to return to work.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 70 years of age.
* Symptomatic primary Great Saphenous Vein "GSV" incompetence diagnosed by clinical symptoms, with or without visible varicosities, and confirmed by duplex ultrasound imaging.
* CEAP classification of C2, C3 or C4.
* Ability to walk unassisted.
* Ability to attend follow-up visits.
* Ability to understand the requirements of the study and to provide written informed consent.
* "GSV" on standing pre-procedure Doppler Ultrasound ≥3mm and ≤10mm (maximum diameter).

Exclusion Criteria:

* Life expectancy < 1 year.
* Regular pain medication.
* Anticoagulation including Heparin or Coumadin.
* Previous Deep Vein Thrombosis "DVT".
* Previous superficial thrombophlebitis in "GSV".
* Previous venous treatment on target limb.
* Known Hyper-coagulable disorder.
* Conditions which prevent routine vein treatment like:

  * Acute disease,
  * Immobilization or inability to ambulate, and
  * Pregnancy.
* Tortuous "GSV", which in the opinion of the Investigator will limit catheter placement. (no 2 primary access sites allowed).
* Incompetent ipsilateral small saphenous or anterior accessory great saphenous vein.
* Known sensitivity to the cyanoacrylate "CA" adhesive.
* Current participation in another clinical study involving an investigational agent or treatment, or within the 30 days prior to enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Comparative Duplex Ultrasound | Immediately Post-procedure
  The Primary endpoint is a change in duplex ultrasound immediately post-procedure as compared to the pre-procedure duplex ultrasound, proving great saphenous vein closure with lack of pathological reflux.

SECONDARY OUTCOMES:
Safety | Immediately post-op through 6 month Follow-up "FU"
  The Secondary endpoint is safety, reflected by the rate of occurrence of all adverse events (procedure and non-procedure related; serious and non-serious).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Proebstle, MD, Principal Investigator — Klinik Proebstlé
Locations (7):
- Aareknudeklinikken, Næstved, Denmark
- Germany (2):
  - Dermatologikum, Hamburg
  - Klinik Proebstle, Mannheim
- Centrum Oosterawal, Alkmaar, Netherlands
- United Kingdom (3):
  - Countess of Chester Hospital NHS Foundation Trust, Chester
  - The Whiteley Clinic, Guildford
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Proebstle T, Alm J, Dimitri S, Rasmussen L, Whiteley M, Lawson J, Davies AH. Three-year follow-up results of the prospective European Multicenter Cohort Study on Cyanoacrylate Embolization for treatment of refluxing great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2021 Mar;9(2):329-334. doi: 10.1016/j.jvsv.2020.05.019. Epub 2020 Jun 26. PMID 32599306
- [Derived] Proebstle TM, Alm J, Dimitri S, Rasmussen L, Whiteley M, Lawson J, Cher D, Davies A. The European multicenter cohort study on cyanoacrylate embolization of refluxing great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2015 Jan;3(1):2-7. doi: 10.1016/j.jvsv.2014.09.001. Epub 2014 Oct 18. PMID 26993674